CLINICAL TRIAL: NCT01275703
Title: Noninvasive Cardiac Output Measurements in Patients With Pulmonary Hypertension Undergoing Exercise Testing
Status: Withdrawn | Type: Observational
Why Stopped: The PI left this institution, and the study was closed.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-180-B
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Pulmonary Hypertension
Keywords: To determine the utility of a noninvasive method of measuring cardiac output during exercise testing in patients with PH
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with PH undergoing exercise testing

SUMMARY:
Subjects in this study have been diagnosed with pulmonary hypertension and their doctors have referred them for an exercise test as part of their normal, routine care. The exercise test will either be a treadmill test or a 6 minute walk test. During a treadmill test, a patient typically walks on a treadmill while their heart is monitored using an electrocardiogram, which records the electrical activity of the heart through 10 small electrode patches attached to the skin of the chest, arms and legs. Additionally, heart rate and blood pressure are monitored throughout the test. A 6-Minute Walk test requires patients to walk for up to 6 minutes to determine how far they can go in order to measure the heart function related to exercise.

The purpose of this study is to measure internal heart pressures using a device called Noninvasive Cardiac Output Monitoring (NICOM) during an exercise test. Normally heart pressures are measured during invasive (meaning that doctors have to go inside the body using a needle or surgery) heart procedures. The NICOM device is non-invasive which means the investigators do not have to go inside the body to obtain the heart pressure measurements. In this study, the investigators will evaluate the non-invasive measurements provided by the NICOM device during the exercise test and see how it relates to information from some of subjects' past heart procedures. This research is being done to devise better, less invasive ways to assess disease severity, track disease progression and evaluate response to therapy.

The NICOM device is approved by the US Food and Drug Administration (FDA) to measure heart pressures. This device is usually used when a patient can't undergo a right heart catheterization. In this study, the investigators are using the device to gather heart pressure measurements for research during the exercise test that is scheduled as part of the subjects' normal, routine care. The research data is being used to devise better, less invasive ways to assess disease severity, track disease progression and evaluate response to therapy. The NICOM device is made by Cheetah Medical.

ELIGIBILITY:
Inclusion Criteria:

* have Pulmonary Hypertension
* undergoing standard of care exercise testing
* 18 years or older

Exclusion Criteria:

* unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 200 consecutive patients referred to the Pulmonary Hypertension Center and scheduled for exercise testing as part of their evaluation of PH.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To determine the utility of a noninvasive method of measuring cardiac output during exercise testing in patients with pulmonary hypertension | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Archer, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States